CLINICAL TRIAL: NCT07164378
Title: Prospective, MulticEnter, Randomized, International Study of the SING IMT™ Prosthesis in Pseudophakic patiEnts With Stable Moderate to Profound Bilateral Central vIsion Impairment Due to adVancEd AMD / PERSPECTIVE Study
Brief Title: International Study of the SING IMT™ Prosthesis in Pseudophakic patiEnts With Stable Moderate to Profound Bilateral Central vIsion Impairment Due to adVancEd AMD / PERSPECTIVE Study
Acronym: PERSPECTIVE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VisionCare, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PKCIP-01.0
Record Dates: First submitted 2025-08-19; First posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Age - Related Macular Degeneration (AMD)
Keywords: Sulcus; AMD; Age-related Macular Degeneration; IOL; Intra-Ocular Lens; Pseudophakic; Samsara Vision; Add-on; SINGIMT; lens-exchange
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lens Exchange group (Experimental): SING IMT™ implantation in the sulcus after removal of the previously implanted IOL
  Interventions: Procedure: Lens-Exchange
- Add-On (Experimental): SING IMT™ implantation in the sulcus in front of an existing IOL
  Interventions: Procedure: Add-on

INTERVENTIONS:
Procedure: Lens-Exchange — The existing IOL will be removed and replaced by implanting SING IMT™ device in the sulcus
  Arms: Lens Exchange group
Procedure: Add-on — The SING IMT™ device will be placed in front of the existing IOL and implanted in the sulcus.
  Arms: Add-On

SUMMARY:
This study aims to expand the CE mark IFU of the SING IMT™ to pseudophakic (patients with an intraocular lents) patients with late stage of AMD (Age-Related Macular Degeneration) and bilateral central vision impairment. This randomized, international, multicenter study will evaluate the safety and efficacy of the device in this patient group. Findings will support regulatory submissions, clinical decision-making, and potential label expansion.

DETAILED DESCRIPTION:
Eligible AMD patients with existing IOL on both eyes will be randomized to either have the SING-IMT device placed on top of the existing IOL, or to replace the existing IOL.

ELIGIBILITY:
Inclusion Criteria:

1. Be 55 years of age or older;
2. Subjects with late-stage AMD; Have retinal findings of geographic atrophy or disciform scar with foveal involvement in both eyes;
3. Had cataract surgery (with IOL implantation in both eyes) at least 6 months prior to enrollment;
4. BCDVA no better than 20/80 and no worse than 20/800 in both eyes.
5. Have adequate peripheral vision in the eye not scheduled for surgery, assessed by observation of ambulation.
6. Achieve using the ETS, at least 2-lines (10 or more letters) improvement in distance on the ETDRS chart in the eye scheduled for surgery.
7. Have an Anterior chambre depth (ACD) of at least 2.5 mm, measured from endothelium, in both eyes.
8. Have an ECD of at least 1600 cells per square mm in both eyes.
9. Be willing to participate in a postoperative training program for the use of the SING IMT™ implant.
10. Review and sign the IEC approved Informed Consent Form (ICF) prior to any clinical investigation-related procedures being performed.
11. Patient is registered with the national social security or equivalent in the country where consent is signed
12. A woman is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies:

13, Not a woman of childbearing potential (WOCBP): A WOCBP who agrees to follow contraceptive guidance starting with the screening visit and through to the end of the study

Exclusion Criteria:

A. Bilateral Ocular Conditions (affecting both eyes):

1. Evidence of active choroidal neovascularization (CNV), or treatment for CNV within the past six (6) months.
2. Diabetic retinopathy.
3. Retinal vascular diseases.
4. History of retinal detachment.
5. Retinitis pigmentosa.
6. Intraocular tumor.
7. Corneal Stromal or Endothelial Dystrophies (for example corneal guttata)Corneal guttata.
8. Patient predisposing to eye rubbing

   B. Surgical Eye Conditions:
9. Narrow angle (i.e., < Schaffer grade 2).
10. Axial length <21 mm or >26 mm.
11. Any history or current ocular or intraocular inflammation, infection, or edema, including but not limited to: - Uveitis, iritis, keratitis, keratouveitis, microbial keratoconjunctivitis.
12. Plate haptic shape IOL implanted.
13. Vitrectomized eye.
14. Zonular weakness, instability, presence of pseudoexfoliation.
15. Iris abnormalities, including but not limited to: Transillumination defects (e.g., pigment dispersion syndrome), aniridia, iris neovascularization.
16. Any IOL already implanted in the sulcus.
17. Presence of toric or multifocal IOL types.
18. Optic Nerve Disease

    C. Systemic or Other General Conditions:
19. A history of steroid-induced IOP elevation uncontrolled, glaucoma, or preoperative IOP >22 mmHg.
20. Known sensitivity to post-operative medications.
21. Significant communication impairment or severe neurological disorders.
22. Administration of any investigational product within 30 days prior to enrolment or planned participation in another clinical investigation during this study.
23. Any condition or situation that, in the opinion of the investigator, may:

    * Put the subject at significant risk,
    * Confound the clinical investigation results, or
    * Interfere significantly with the subject's participation in the study.
24. Individuals under legal care (e.g., incarcerated patients or those under legal guardianship) who are unable to understand and provide informed consent.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2025-09-30 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
percentage of ECD loss | at baseline, then at 1, 3 and 6 months
  assessed within each treatment group relative to baseline (pre-surgery). The ECD loss should not exceed 23%

SECONDARY OUTCOMES:
Incision size required for device implantation | baseline
  measurement of the incision size
Number of Surgical Complications, AEs and SAEs | at baseline, then at 1, 3 and 6 months
  Assess number of safety events comparing to similar procedures.
Acuity | at baseline, then at 1, 3 and 6 months
  Change in near and distance best corrected acuity in implanted eyes
Patient-reported outcomes | at baseline, then at 1, 3 and 6 months
  Using the Impact of Vision Impairment (IVI) questionnaire, 28 questions are answered, providing 4 different scores:
  1. Vision-related quality of life Average of all items (ranging from 0 to 2.9)
  2. Reading and accessing information Average of (Q1, Q3, Q5, Q6, Q7, Q8, Q9, Q14, Q15), (ranging from 0 to 2.7)
  3. Mobility and Independence Average of (Q2, Q4, Q10, Q11, Q12, Q13, Q16, Q17, Q18, Q19, Q20), (ranging from 0 to 3)
  4. Emotional well-being Average of (Q21, Q22, Q23, Q24, Q25, Q26, Q27, Q28), (ranging from 0 to 3)

CONTACTS AND LOCATIONS:
Locations (11):
- France (3):
  - Centre d'Ophtalmologie Paradis-Monticelli, Marseille
  - Hélios Ophtalmologie, Saint-Jean-de-Luz
  - CHU de Strasbourg, Strasbourg
- Germany (3):
  - Asklepios Augenklinik Nord-Heidberg, Hamburg
  - Augenklinik Sulzbach, Sulzbach
  - Augenklinik und Poliklinik des Universitätsklinikums, Würzburg
- Italy (5):
  - Ospedale Generale Regionale "F. Miulli", Bari
  - IRCCS Humanitas, Bergamo
  - Azienda Ospedaliero-Universitaria di Ferrara, Ferrara
  - Presidio Ospedaliero Palagi, Florence
  - Policlinico Universitario Fondazione Agostino Gemelli, Roma

IPD SHARING:
Plan to Share IPD: No